CLINICAL TRIAL: NCT02473289
Title: A Double-Blind, Placebo-Controlled, Multicenter Study of Sirukumab as Adjunctive Treatment to a Monoaminergic Antidepressant in Adults With Major Depressive Disorder
Brief Title: An Efficacy and Safety Study of Sirukumab in Participants With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107171; CNTO136MDD2001 (Other: Janssen Research & Development, LLC); 2014-005206-37 (EudraCT Number)
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive disorder, major; Sirukumab
MeSH Terms: conditions — Depressive Disorder, Major | interventions — sirukumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Sirukumab 50 milligram (mg) (Experimental): Participants will receive sirukumab 50 mg as subcutaneous injection on Day 1, 28 and 56.
  Interventions: Drug: Sirukumab 50 mg
- Placebo (Placebo Comparator): Participants will receive matching placebo on Day 1, 28 and 56.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sirukumab 50 mg — Participants will receive sirukumab 50 mg as subcutaneous injection on Day 1, 28 and 56.
  Arms: Sirukumab 50 milligram (mg)
Drug: Placebo — Participants will receive matching placebo on Day 1, 28 and 56.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of sirukumab as adjunctive treatment to antidepressant therapy (monoaminergic antidepressant) where sirukumab (administered as a 50 milligram (mg) subcutaneous (SC) injection at Day 1, Day 28 and Day 56 during the 12- week double-blind treatment period) is compared to adjunctive placebo based on the change from baseline to 12-week endpoint in depressive symptoms as measured by the total score on the Hamilton Depression Rating Scale (HDRS), in participants diagnosed with Major Depressive Disorder (MDD) who have had a suboptimal response to the current standard oral antidepressant therapy and have a screening high sensitivity C-Reactive Protein (hsCRP) >=0.300 milligram per deciliters (mg/dL) (International System of Units (SI) 3.00 mg/L). A cohort of subjects with hsCRP <0.300 milligram per deciliter will also be enrolled to allow a better understanding of the relationship between CRP and clinical changes.

DETAILED DESCRIPTION:
A double-blind, placebo-controlled, multicenter study of sirukumab as adjunctive treatment to a monoaminergic antidepressant in adults with major depressive disorder. Participants will be randomly assigned to receive either placebo or sirukumab 50 milligram (mg) at a ratio of 1:1 at Day 1, 28 and 56. Participants will primarily be assessed for change from baseline in Hamilton Depression Rating Scale (HDRS17) score at Week 12. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a primary DSM-5 diagnosis of MDD
* Must have a HDRS total score greater than or equal to (>=) 18 at screening and predose at Day 1, as recorded by the remote independent rater and must not demonstrate an improvement of > 25 percent (%) on their HDRS total score from the screening to baseline visit
* Must be medically stable on the basis of physical examination, medical history, vital signs, clinical laboratory tests and 12-lead ECG performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the subject's source documents and initialed by the investigator
* Participants with hypothyroidism who are on stable treatment for 3 months prior to screening are required to have thyroid stimulating hormone (TSH) and free thyroxine (FT4) obtained. If the TSH value is out of range, but FT4 is normal, such cases should be discussed directly with the medical monitor before the subject is enrolled. If the FT4 value is out of range, the participant is not eligible

Exclusion Criteria:

* Any other current Axis one psychiatric condition, including, but not limited to, MDD with current psychotic features, bipolar disorder (including lifetime diagnosis), obsessive-compulsive disorder, borderline personality disorder, eating disorder (eg, bulimia, anorexia nervosa), or schizophrenia (lifetime). The MINI will be used to screen for comorbid psychiatric diagnoses. As noted above, subjects with a diagnosis of comorbid GAD, Post-Traumatic Stress Disorder, Persistent Depressive Disorder, ADHD, Social Anxiety Disorder, Panic Disorder with or without agoraphobia or Nicotine/Caffeine Dependence may be included, if the investigator considers MDD to be the primary diagnosis
* A history of alcohol or substance use disorder (abuse/dependence) within 6 months prior to screening (nicotine and caffeine dependence are not exclusionary)
* A current or recent (within the past year) history of clinically significant suicidal ideation (corresponding to a score of >= 3 for ideation) or any suicidal behavior within the past year, as validated on the C-SSRS at screening or baseline. Subjects with a prior suicide attempt of any sort, or history of prior serious suicidal ideation/plan should be carefully screened for current suicidal ideation and only included at the discretion of the investigator
* More than 3 failed antidepressant treatments (of adequate dose and duration) in the current episode of depression (verified by the MGH-ATRQ)
* Length of current major depressive episode > 60 months

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 193 (Actual)
Dates: Start 2015-07-23 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (46):
- United States (24):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Bellflower, California
  - Glendale, California
  - Lemon Grove, California
  - Orange, California
  - Santa Ana, California
  - Torrance, California
  - Wildomar, California
  - Atlanta, Georgia
  - Decatur, Georgia
  - Chicago, Illinois
  - Edgewood, Kentucky
  - Baltimore, Maryland
  - Grand Rapids, Michigan
  - Lebanon, New Hampshire
  - Brooklyn, New York
  - New York, New York
  - Staten Island, New York
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Houston, Texas
  - Plano, Texas
  - Salt Lake City, Utah
- Canada (4):
  - Edmonton, Alberta
  - Chatham, Ontario
  - Hamilton, Ontario
  - Toronto, Ontario
- Poland (5):
  - Bełchatów
  - Bydgoszcz
  - Chełmno
  - Gorlice
  - Lublin
- Russia (9):
  - Karelia
  - Moscow
  - Nizny Novgorod
  - Rostov-on-Don
  - Saint Petersburg
  - Saratov
  - Saratov Region
  - Tomsk
  - Yaroslavl
- United Kingdom (4):
  - Edinburgh
  - Glasgow
  - Oxford
  - Redruth

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo subcutaneous (SC) injection on Day 1, Day 28 and Day 56, while continuing their baseline oral monoaminergic antidepressant(s).
- Sirukumab 50 mg: Participants received sirukumab 50 milligram (mg) on Day 1, Day 28 and Day 56, while continuing their baseline oral monoaminergic antidepressant(s).
Period: Overall Study
Arm/Group | Placebo | Sirukumab 50 mg
Started | 99 | 94
Completed | 88 | 81
Not Completed | 11 | 13
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal of consent | 6 | 7
Not completed — Treatment Unblinded + Adverse event | 0 | 1
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sirukumab 50 mg | Total
Number analyzed (Participants) | 99 | 94 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (11.73) | 45.4 (10.83) | 44.7 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 74 | 149
  Male | 24 | 20 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 95 | 89 | 184
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 5 | 15
  White | 86 | 87 | 173
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black or African American | 10 | 5 | 15
  Hispanic or Latino | 4 | 4 | 8
  Other | 2 | 1 | 3
  White Non-Hispanic | 82 | 83 | 165
Region of Enrollment [Count of Participants; unit: Participants]
  CANADA | 5 | 2 | 7
  POLAND | 21 | 19 | 40
  RUSSIAN FEDERATION | 48 | 47 | 95
  UNITED KINGDOM | 2 | 1 | 3
  UNITED STATES | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Depression Rating Scale (HDRS-17) Total Score at Week 12
Description: The HDRS-17 is a clinician-administered rating scale designed to assess the severity of symptoms in participants diagnosed with depression with a score range of 0 to 52. Each of the 17 items is rated by the clinician on either a 3-point (0 to 2) or a 5-point scale (0 to 4). The point scale used a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). A total score (0 to 52) was calculated by adding the scores of all 17 items. For each item as well as the total score, a higher score represents a more severe condition. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Time Frame: Baseline and Week 12
Population: Modified Intent-to-treat 1 (mITT1) analysis set: all randomized participants with high sensitivity c-reactive protein (hsCRP) >= 3.00 milligram per liter (mg/L) at screening and baseline who receive at least 1 dose of study drug and have both baseline and at least one postbaseline HDRS-17 total score in double-blind (DB) treatment period.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Sirukumab 50 mg
Number analyzed (Participants) | 42 | 44
Units on a scale | -10.6 (1.43) | -11.4 (1.52)
Statistical Analysis 1: Comparison: Placebo vs Sirukumab 50 mg; Test type: Superiority; p = 0.310, MMRM — 1-sided; Here 'MMRM' refers to Mixed-effect Model Using Repeated Measures; Difference of Least Square (LS) Means = -0.8, 75% CI 2-sided [-2.77 to 1.10], Standard Error of Mean 1.67

2. Secondary Outcome: Change From Baseline in HDRS-17 Total Score at Weeks 1, 4 and 8
Description: The HDRS-17 is a clinician-administered rating scale designed to assess the severity of symptoms in participants diagnosed with depression with a score range of 0 to 52. Each of the 17 items is rated by the clinician on either a 3-point (0 to 2) or a 5-point scale (0 to 4). The point scale used a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). A total score (0 to 52) was calculated by adding the scores of all 17 items. For each item as well as the total score, a higher score represents a more severe condition.
Time Frame: Baseline, Weeks 1, 4 and 8
Population: mITT1 analysis set: all randomized participants with hsCRP >= 3.00 mg/L at screening and baseline who receive at least 1 dose of study drug and have both baseline and at least one postbaseline HDRS-17 total score in DB treatment period. 'n' (number of participants analyzed)- number of participants analyzed at each specified timepoint, for each arm.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Sirukumab 50 mg
Number analyzed (Participants) | 47 | 47
Units on a scale
  Change at Week 1: number analyzed (Participants) | 46 | 47
  Change at Week 1 | -5.1 (1.03) | -4.6 (1.15)
  Change at Week 4: number analyzed (Participants) | 46 | 45
  Change at Week 4 | -7.5 (1.21) | -7.8 (1.33)
  Change at Week 8: number analyzed (Participants) | 42 | 45
  Change at Week 8 | -7.9 (1.29) | -11.0 (1.39)

3. Secondary Outcome: Percentage of Participants With Remission as Assessed by HDRS-17 Total Score at Week 12
Description: Remission- Percentage of participants with HDRS-17 total score less than or equal to (<=) 7 were considered as remitters. HDRS-17 defined as clinician-administered rating scale designed to assess severity of symptoms in participants diagnosed with depression with score range of 0 to 52. Each of 17 items is rated by clinician on either a 3-point (0 to 2) or a 5-point scale (0 to 4). The point scale used a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). A total score (0 to 52) was calculated by adding scores of all 17 items. For each item as well as total score, a higher score represents a more severe condition.
Time Frame: Week 12
Population: mITT1 analysis set: all randomized participants with hsCRP >=3.00 mg/L at screening and baseline who receive at least 1 dose of study drug and have both baseline and at least one postbaseline HDRS-17 total score in DB treatment period. 'N' (number of participants analyzed)- number of participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Sirukumab 50 mg
Number analyzed (Participants) | 42 | 44
Percentage of participants | 19.0 | 15.9

4. Secondary Outcome: Percentage of Participants With Response as Assessed by HDRS-17 Total Score at Week 12
Description: Response- Percentage of participants with greater than or equal to (>=) 50 percent (%) improvement on the HDRS-17 total score from baseline at Week 12 were considered as responders. The HDRS-17 defined as clinician-administered rating scale designed to assess the severity of symptoms in participants diagnosed with depression with a score range of 0 to 52. Each of the 17 items is rated by the clinician on either a 3-point (0 to 2) or a 5-point scale (0 to 4). The point scale used a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). A total score (0 to 52) was calculated by adding the scores of all 17 items. For each item as well as the total score, a higher score represents a more severe condition.
Time Frame: Week 12
Population: mITT1 analysis set: all randomized participants with hsCRP >= 3.00 mg/L at screening and baseline who receive at least 1 dose of study drug and have both baseline and at least one postbaseline HDRS-17 total score in DB treatment period. 'N' (number of participants analyzed)- number of participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Sirukumab 50 mg
Number analyzed (Participants) | 42 | 44
Percentage of participants | 33.3 | 34.1

5. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Total Score at Weeks 1, 4, 8, 12, 16, and 22
Description: CGI-S defined as clinician-rated scale that assesses the severity of mental illness on a scale of 0 to 7. Considering total clinical experience, a participant was assessed on severity of mental illness at the time of rating according to:1: normal, not at all ill; 2: borderline mentally ill; 3: mildly ill; 4: moderately ill; 5: markedly ill; 6: severely ill; 7: among the most extremely ill patients. A higher score implies a more severe condition.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, and 22
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Sirukumab 50 mg
Number analyzed (Participants) | 47 | 47
Units on a scale
  Change at Week 1: number analyzed (Participants) | 46 | 47
  Change at Week 1 | -0.6 (0.14) | -0.7 (0.15)
  Change at Week 4: number analyzed (Participants) | 46 | 45
  Change at Week 4 | -1.1 (0.16) | -1.0 (0.17)
  Change at Week 8: number analyzed (Participants) | 42 | 45
  Change at Week 8 | -1.4 (0.18) | -1.5 (0.19)
  Change at Week 12: number analyzed (Participants) | 44 | 44
  Change at Week 12 | -1.5 (0.21) | -1.9 (0.22)
  Change at Week 16: number analyzed (Participants) | 42 | 44
  Change at Week 16 | -1.9 (0.23) | -2.1 (0.24)
  Change at Week 22: number analyzed (Participants) | 42 | 43
  Change at Week 22 | -2.0 (0.24) | -2.3 (0.25)

6. Secondary Outcome: Change From Baseline in Patient Health Questionnaire (PHQ-9) Total Score at Weeks 1, 4, 8, 12, 16, and 22
Description: The PHQ-9 used as a participant-reported measure of depressive symptomatology. The PHQ-9 is 9-item scale, where each item is rated on a 4-point scale (0=Not at all, 1=Several Days, 2=More than half the days, and 3=Nearly every day). The participant's item responses were summed to provide a total score range of 0 to 27. Higher scores indicates greater severity of depressive symptoms. The recall period is 2 weeks.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, and 22
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Sirukumab 50 mg
Number analyzed (Participants) | 47 | 47
Units on a scale
  Change at Week 1: number analyzed (Participants) | 45 | 47
  Change at Week 1 | -2.5 (0.58) | -3.1 (0.61)
  Change at Week 4: number analyzed (Participants) | 45 | 45
  Change at Week 4 | -4.4 (0.75) | -5.3 (0.79)
  Change at Week 8: number analyzed (Participants) | 41 | 45
  Change at Week 8 | -5.6 (0.86) | -7.6 (0.87)
  Change at Week 12: number analyzed (Participants) | 43 | 44
  Change at Week 12 | -7.5 (0.98) | -8.9 (1.00)
  Change at Week 16: number analyzed (Participants) | 42 | 44
  Change at Week 16 | -8.2 (0.98) | -9.6 (1.00)
  Change at Week 22: number analyzed (Participants) | 41 | 43
  Change at Week 22 | -9.1 (1.04) | -10.7 (1.05)

7. Secondary Outcome: Change From Baseline in Snaith Hamilton Pleasure Scale (SHAPS) Total Score (Definition 1) at Weeks 1, 4, 8, 12, 16, and 22
Description: The Snaith-Hamilton Pleasure Scale (SHAPS) is short, 14-item instrument to measure anhedonia. Each of the 14 items has a set of four response categories (Definition 1): Definitely Agree (=1), Agree (= 2), Disagree (= 3), and Definitely Disagree (= 4). A SHAPS total score was calculated as the sum of the 14 item scores with a total score range from 14 to 56. A higher total score indicates higher levels of state anhedonia.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, and 22
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Sirukumab 50 mg
Number analyzed (Participants) | 47 | 47
Units on a scale
  Change at Week 1: number analyzed (Participants) | 45 | 47
  Change at Week 1 | -1.4 (0.72) | -3.3 (0.74)
  Change at Week 4: number analyzed (Participants) | 45 | 45
  Change at Week 4 | -3.9 (0.75) | -5.1 (0.78)
  Change at Week 8: number analyzed (Participants) | 41 | 45
  Change at Week 8 | -5.8 (0.87) | -7.0 (0.88)
  Change at Week 12: number analyzed (Participants) | 43 | 44
  Change at Week 12 | -5.9 (1.00) | -8.9 (1.02)
  Change at Week 16: number analyzed (Participants) | 42 | 44
  Change at Week 16 | -7.0 (1.11) | -8.8 (1.12)
  Change at Week 22: number analyzed (Participants) | 41 | 43
  Change at Week 22 | -7.8 (1.11) | -10.6 (1.12)

8. Secondary Outcome: Change From Baseline in Snaith Hamilton Pleasure Scale (SHAPS) Total Score (Definition 2) at Weeks 1, 4, 8, 12, 16, and 22
Description: The Snaith-Hamilton Pleasure Scale (SHAPS) is short, 14-item instrument to measure anhedonia. Each of the 14 items has a set of four response categories (Definition 2): Definitely Agree (= 0), Agree (= 0), Disagree (= 1), and Definitely Disagree (= 1). A SHAPS total score was calculated as the sum of the 14 item scores with a score range from 0 to 14. A higher total score indicates higher levels of state anhedonia.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, and 22
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Sirukumab 50 mg
Number analyzed (Participants) | 47 | 47
Units on a scale
  Change at Week 1: number analyzed (Participants) | 45 | 47
  Change at Week 1 | -1.2 (0.45) | -2.0 (0.47)
  Change at Week 4: number analyzed (Participants) | 45 | 45
  Change at Week 4 | -2.2 (0.49) | -3.3 (0.51)
  Change at Week 8: number analyzed (Participants) | 41 | 45
  Change at Week 8 | -3.6 (0.57) | -4.4 (0.57)
  Change at Week 12: number analyzed (Participants) | 43 | 44
  Change at Week 12 | -3.7 (0.64) | -5.4 (0.66)
  Change at Week 16: number analyzed (Participants) | 42 | 44
  Change at Week 16 | -4.1 (0.69) | -5.6 (0.70)
  Change at Week 22: number analyzed (Participants) | 41 | 43
  Change at Week 22 | -4.6 (0.71) | -6.8 (0.72)

9. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Total Score at Weeks 1, 4, 8, 12, 16, and 22
Description: The FACIT-Fatigue is a questionnaire that assesses self-reported tiredness, weakness, and difficulty conducting usual activities due to fatigue. The subscale consists 13-item instrument to measure fatigue. Each of the 13 items has a set of five response categories: Not at all (=0), A little bit (=1), Somewhat (=2), Quite a bit (=3) and Very much (=4). A total FACIT-Fatigue subscale score was calculated as the sum of the 13 item scores (reserved scores [4 - score] for all except for 2 items: "I have energy" and "I am able to do my usual activities"), and ranges from 0 to 52, with a higher score indicating less fatigue.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, and 22
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Sirukumab 50 mg
Number analyzed (Participants) | 47 | 47
Units on a scale
  Change at Week 1: number analyzed (Participants) | 45 | 47
  Change at Week 1 | 1.75 (4.671) | 4.91 (10.097)
  Change at Week 4: number analyzed (Participants) | 45 | 45
  Change at Week 4 | 6.87 (10.119) | 6.44 (9.633)
  Change at Week 8: number analyzed (Participants) | 41 | 45
  Change at Week 8 | 8.93 (9.913) | 10.09 (10.346)
  Change at Week 12: number analyzed (Participants) | 43 | 44
  Change at Week 12 | 11.65 (13.476) | 13.82 (11.486)
  Change at Week 16: number analyzed (Participants) | 42 | 44
  Change at Week 16 | 13.55 (12.029) | 13.95 (12.066)
  Change at Week 22: number analyzed (Participants) | 41 | 43
  Change at Week 22 | 14.54 (13.585) | 17.23 (12.051)

ADVERSE EVENTS:
Time Frame: Approximately 26 weeks
Arm/Group | Placebo | Sirukumab 50 mg
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/94
Serious Adverse Events (participants affected / at risk) | 2/99 | 3/94
Other Adverse Events (participants affected / at risk) | 13/99 | 19/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=99) | Sirukumab 50 mg (N=94)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Transaminases Increased (Investigations) | 1 | 0
Depression Suicidal (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=99) | Sirukumab 50 mg (N=94)
Injection Site Erythema (General disorders) | 0 | 11
Injection Site Pain (General disorders) | 1 | 5
Headache (Nervous system disorders) | 12 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT02473289/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT02473289/SAP_001.pdf